CLINICAL TRIAL: NCT02027428
Title: A Phase III, Randomized, Open-Label, Multi-Center, Safety and Efficacy Study to Evaluate Nab-Paclitaxel (Abraxane®) as Maintenance Treatment After Induction With Nab-Paclitaxel Plus Carboplatin in Subjects With Squamous Cell Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety and Efficacy Study of Abraxane as Maintenance Treatment After Abraxane Plus Carboplatin in 1st Line Stage IIIB / IV Squamous Cell Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-NSCL-003; 2014-003804-66 (EudraCT Number)
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Squamous Cell Carcinoma, Non-Small-Cell Lung
Keywords: Nab-paclitaxel; Albumin bound paclitaxel; Taxanes; Maintenance trials; Celgene; Abraxane; ABI-007; NSCLC; Non-Small Cell Lung Cancer; Cancer of the Lung; Carcinoma, Squamous Cell; Lung Neoplasms; Abound.sqm
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Albumin-Bound Paclitaxel; Neoadjuvant Therapy; 130-nm albumin-bound paclitaxel; Carboplatin; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abraxane + Best Supportive Care (BSC) (Experimental): Dosing will occur in two phases - induction and maintenance. During induction, the subject will receive Abraxane plus carboplatin as standard of care. At the end of 4 cycles, if the subject has a complete response, partial response, or stable disease, he/she will continue on to the maintenance phase. Maintenance dosing on this arm includes Abraxane plus best supportive care.
  Interventions: Drug: Abraxane (Induction); Drug: Carboplatin (Induction); Drug: Abraxane (Maintenance); Other: Best Supportive Care (Maintenance)
- Best Supportive Care (BSC) (Other): Dosing will occur in two phases - induction and maintenance. During induction, the subject will receive Abraxane plus carboplatin as standard of care. At the end of 4 cycles, if the subject has a complete response, partial response, or stable disease, he/she will continue on to the maintenance phase. Maintenance dosing on this arm includes best supportive care only.
  Interventions: Drug: Abraxane (Induction); Drug: Carboplatin (Induction); Other: Best Supportive Care (Maintenance)

INTERVENTIONS:
Drug: Abraxane (Induction) — 100 mg/m2 IV infusion over 30 minutes on Days 1 and 8 and 15 of each 21-day cycle, administered as standard of care
  Other Names: nab-paclitaxel
  Arms: Abraxane + Best Supportive Care (BSC)
Drug: Carboplatin (Induction) — 6 mg/min/mL IV on Day 1 of each 21-day cycle after completion of nab-paclitaxel infusion
  Arms: Abraxane + Best Supportive Care (BSC)
Drug: Abraxane (Maintenance) — 100 mg/m2 IV infusion over 30 minutes on Days 1 and 8 of each 21-day cycle, administered as standard of care
  Arms: Abraxane + Best Supportive Care (BSC)
Other: Best Supportive Care (Maintenance) — The best palliative care per investigator (including but not limited to: antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, nutritional support, and/or focal external-beam radiation for control of pain, cough, dyspnea, or hemoptysis), excluding antineoplastic agents
  Arms: Abraxane + Best Supportive Care (BSC)
Drug: Abraxane (Induction) — 100 mg/m2 IV infusion over 30 minutes on Days 1 and 8 and 15 of each 21-day cycle, administered as standard of care
  Other Names: nab-paclitaxel
  Arms: Best Supportive Care (BSC)
Drug: Carboplatin (Induction) — 6 mg/min/mL IV on Day 1 of each 21-day cycle after completion of nab-paclitaxel infusion, administered as standard of care
  Arms: Best Supportive Care (BSC)
Other: Best Supportive Care (Maintenance) — The best palliative care per investigator (including but not limited to: antibiotics, analgesics, antiemetics, thoracentesis, pleurodesis, blood transfusions, nutritional support, and/or focal external-beam radiation for control of pain, cough, dyspnea, or hemoptysis), excluding antineoplastic agents
  Arms: Best Supportive Care (BSC)

SUMMARY:
Maintenance treatment of advanced stage squamous cell NSCLC.

Phase III, randomized, open-label, multi-center study of nab-paclitaxel with best supportive care (BSC) or BSC alone as maintenance treatment after response or stable disease (SD) with nab-paclitaxel plus carboplatin as induction in subjects with stage IIIB/IV squamous cell NSCLC.

Subjects who discontinued treatment from the maintenance part for any reason other than withdrawal of consent, lost to follow-up, or death, were entered into a Follow-up period that had a visit 28 days after progression or discontinuation.

Those who entered Follow-up without progression continued with follow-up scans according to standard of care (SOC) until documentation of progression of disease. Additionally, subjects were followed for OS by phone approximately every 90 days for a minimum of 18 months, for up to approximately 5 years after the last subject was randomized.

DETAILED DESCRIPTION:
The sponsor used 15 Sep 2017 as the database cut-off date.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age at the time of signing the Informed Consent Form.
2. Understand and voluntarily provide written consent to the Informed Consent Form prior to conducting any study related assessments/procedures.
3. Able to adhere to the study visit schedule and other protocol requirements

   Disease Specific
4. Histologically or cytologically confirmed Stage IIIB or IV squamous cell Non Small Cell Lung Cancer at study entry.
5. No other current active malignancy requiring anticancer therapy.
6. Radiographically documented measurable disease at study entry (as defined by the Response Evaluation Criteria In Solid Tumors [RECIST] v1.1 criteria).
7. No prior chemotherapy for the treatment of metastatic disease at study entry. Adjuvant chemotherapy is permitted providing cytotoxic chemotherapy was completed 12 months prior to starting the study and without disease recurrence.
8. Absolute neutrophil count ≥ 1500 cells/mm^3.
9. Platelets ≥ 100,000 cells/mm^3.
10. Hemoglobin ≥ 9 g/dL.
11. Aspartate transaminase/serum glutamic oxaloacetic transaminase, alanine transaminase/serum glutamic pyruvic transaminase ≤ 2.5 × upper limit of normal range or ≤ 5.0 × upper limit of normal range if liver metastases.
12. Total bilirubin ≤ 1.5 × upper limit of normal range except in cases of Gilbert's disease and liver metastases.
13. Creatinine ≤ 1.5 mg/dL.
14. Expected survival of > 12 weeks for the Induction part of the study.
15. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
16. For Maintenance part of the study, subjects must have received at least one dose of nab-paclitaxel in each of the 4 cycles during Induction

    Pregnancy
17. Females of childbearing potential [defined as a sexually mature woman who (1) have not undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or (2) have not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months)] must:

    1. agree to take a pregnancy test prior to starting study medication and throughout the study participation.
    2. commit to complete abstinence from heterosexual contact, or agree to use medical doctor-approved contraception throughout the study without interruption, and while receiving study medication or for a longer period if required by local regulations.
18. Male subjects must:

    c. agree to complete abstinence from heterosexual contact or use a condom during sexual contact with a female of child bearing potential while receiving study medication and within 6 months after last dose of study medication, even if he has undergone a successful vasectomy.
19. Females must abstain from breastfeeding during study participation and 3 months after IP discontinuation.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment into the Induction and Maintenance parts of the study (except if specified at study entry only):

1. Evidence of active brain metastases, including leptomeningeal involvement (prior evidence of brain metastasis are permitted only if treated and stable and off therapy for ≥ 4 weeks prior to first dose of study drug).
2. Only evidence of disease is non-measurable at study entry.
3. Preexisting peripheral neuropathy of Grade 2, 3, or 4 (per Common Terminology Criteria for Adverse Events v4.0).
4. Venous thromboembolism within 6 months prior to signing Informed Consent Form.
5. Current congestive heart failure (New York Heart Association class II-IV).
6. History of the following within 6 months prior to first administration of a study drug: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant electrocardiogram (ECG) abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder.
7. Treatment with any investigational product within 28 days prior to signing Informed Consent Form.
8. History of allergy or hypersensitivity to nab-paclitaxel or carboplatin.
9. Currently enrolled in any other clinical protocol or investigational trial that involved administration of experimental therapy and/or therapeutic devices.
10. Any other clinically significant medical condition and/or organ dysfunction that will interfere with the administration of the therapy according to this protocol.
11. Subject has any other malignancy within 5 years prior to randomization. Exceptions include the following: squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, uteri, non-melanomatous skin cancer, carcinoma in situ of the breast, or incidental histological finding of prostate cancer (TNM stage of T1a or T1b) - all treatments that should have been completed 6 months prior to signing informed consent form (ICF).
12. Subject has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting investigational product (IP), and/or from whom ≥ 30% of the bone marrow was irradiated. Prior radiation therapy to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed.
13. Pregnant and nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teng Jin Ong, MD, Study Director — Celgene
Locations (119):
- United States (91):
  - Clearview Cancer Institute Oncology Specialties, P.C, Huntsville, Alabama
  - Palo Verde Hematology Oncology, Ltd., Glendale, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - City of Hope Cancer Center, Duarte, California
  - Cancer Care Associates of Fresno Medical Group Inc, Fresno, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Clinical Trials and Research Associates, Montebello, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Lynn Cancer Institute, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic, LLP Center for Cancer Care and Research, Lakeland, Florida
  - University of Miami Miller School of Medicine Jackson Memorial Hospital, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Memorial Cancer Institute West, Pembroke Pines, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University Cancer and Blood Center, LLC, Athens, Georgia
  - University of Chicago, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Kansas University Medical Center, Westwood, Kansas
  - Cancer Center of Kansas (MAT), Wichita, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville, J.G. Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute Louisville Oncology, Louisville, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Eastern Maine Medical Center, Brewer, Maine
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Western Michigan Cancer Center, Kalamazoo, Michigan
  - St Joseph Oncology, Saint Joseph, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hematology-Oncology Associates of NNJ, P, Morristown, New Jersey
  - New York Oncology Hematology P.C., Albany, New York
  - Clinical Research Alliance, Lake Success, New York
  - NYU Langone Medical Center, Lake Success, New York
  - Beth Israel Medical Centers, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Montefiore Medical Center Albert Einstein Cancer Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Moses H. Cone Regional Cancer Center, Greensboro, North Carolina
  - Hematology and Oncology Associates, Inc., Canton, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Mark H. Zangmeister Center, Columbus, Ohio
  - Tri-County Hematology and Oncology Associates, Massillon, Ohio
  - Toledo Community Oncology Program, Toledo, Ohio
  - Mercy Clinic Oklahoma Communities, Inc., Oklahoma City, Oklahoma
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Erie Regional Cancer Center, Erie, Pennsylvania
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center - Cancer Pavilion, Pittsburgh, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Chattanooga Oncology Hematology Care, Chattanooga, Tennessee
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - TX Onc, PA- Beaumont, Beaumont, Texas
  - Brooke Army Medical Center Francis Street Medical Center, Fort Sam Houston, Texas
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - UT Health Oncology, Houston, Texas
  - Millenium Oncology, Houston, Texas
  - TX Onc Tyler Cancer Center, Tyler, Texas
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - St Mary's Medical Center, Huntington, West Virginia
  - West Virginia University, Berkeley Medical Center, Cancer and Infusion Center, Martinsburg, West Virginia
  - West Virginia University, Berkeley Medical Center, Cancer and Infusion Center, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (10):
  - Kliniken der Stadt Koln gGmbH - Krankenhaus Merheim, Cologne
  - St. Antonius Hospital, Eschweiler
  - Asklepios Fachkliniken Muenchen Gauting, Gauting
  - Universitatsklinikum Halle Saale, Halle
  - Diakoniekrankenhaus Halle, Halle
  - Thorax Klinik, Heidelberg
  - Universitat Des Saarlandes, Homburg
  - Lungenklinik Lostau gGmbH, Lostau
  - Klinik Loewenstein gGmbH, Löwenstein
  - Universitatsklinikum Ulm, Ulm
- Italy (8):
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialita San Giuseppe Moscati, Avellino
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S.Orsola Malpighi, Bologna
  - Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona
  - Istituto Nazionale Per La Ricerca Sul Cancro, Genova
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Istituto Nazionale Tumori Regina Elena di Roma, Roma
  - Ospedale San Vincenzo Taormina, Taormina
- Spain (8):
  - Intituto Catalán de Oncología de Girona, Girona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Lozano Blesa, Zaragoza
- United Kingdom (2):
  - Churchhill Hospital, Oxford
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Background] Thomas M, Spigel DR, Jotte RM, McCleod M, Socinski MA, Page RD, Gressot L, Knoble J, Juan O, Morgensztern D, Isla D, Kim ES, West H, Ko A, Ong TJ, Trunova N, Gridelli C. nab-paclitaxel/carboplatin induction in squamous NSCLC: longitudinal quality of life while on chemotherapy. Lung Cancer (Auckl). 2017 Oct 30;8:207-216. doi: 10.2147/LCTT.S138570. eCollection 2017. PMID 29138610
- [Background] Mudad R, Patel MB, Margunato-Debay S, Garofalo D, Lal LS. Comparative effectiveness and safety of nab-paclitaxel plus carboplatin vs gemcitabine plus carboplatin in first-line treatment of advanced squamous cell non-small cell lung cancer in a US community oncology setting. Lung Cancer (Auckl). 2017 Oct 19;8:179-190. doi: 10.2147/LCTT.S139647. eCollection 2017. PMID 29089791
- [Background] Reni M, Zanon S, Balzano G, Passoni P, Pircher C, Chiaravalli M, Fugazza C, Ceraulo D, Nicoletti R, Arcidiacono PG, Macchini M, Peretti U, Castoldi R, Doglioni C, Falconi M, Partelli S, Gianni L. A randomised phase 2 trial of nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in locally advanced or borderline resectable pancreatic adenocarcinoma. Eur J Cancer. 2018 Oct;102:95-102. doi: 10.1016/j.ejca.2018.07.007. Epub 2018 Aug 24. PMID 30149366
- [Background] Yardley DA, Coleman R, Conte P, Cortes J, Brufsky A, Shtivelband M, Young R, Bengala C, Ali H, Eakel J, Schneeweiss A, de la Cruz-Merino L, Wilks S, O'Shaughnessy J, Gluck S, Li H, Miller J, Barton D, Harbeck N; tnAcity investigators. nab-Paclitaxel plus carboplatin or gemcitabine versus gemcitabine plus carboplatin as first-line treatment of patients with triple-negative metastatic breast cancer: results from the tnAcity trial. Ann Oncol. 2018 Aug 1;29(8):1763-1770. doi: 10.1093/annonc/mdy201. PMID 29878040
- [Background] Ailawadhi S, DerSarkissian M, Duh MS, Lafeuille MH, Posner G, Ralston S, Zagadailov E, Ba-Mancini A, Rifkin R. Cost Offsets in the Treatment Journeys of Patients With Relapsed/Refractory Multiple Myeloma. Clin Ther. 2019 Mar;41(3):477-493.e7. doi: 10.1016/j.clinthera.2019.01.009. Epub 2019 Feb 14. PMID 30773308
- [Background] Kim S, Signorovitch JE, Yang H, Patterson-Lomba O, Xiang CQ, Ung B, Parisi M, Marshall JL. Comparative Effectiveness of nab-Paclitaxel Plus Gemcitabine vs FOLFIRINOX in Metastatic Pancreatic Cancer: A Retrospective Nationwide Chart Review in the United States. Adv Ther. 2018 Oct;35(10):1564-1577. doi: 10.1007/s12325-018-0784-z. Epub 2018 Sep 12. PMID 30209750
- [Background] Weiss J, Gilbert J, Deal AM, Weissler M, Hilliard C, Chera B, Murphy B, Hackman T, Liao JJ, Grilley Olson J, Hayes DN. Induction chemotherapy with carboplatin, nab-paclitaxel and cetuximab for at least N2b nodal status or surgically unresectable squamous cell carcinoma of the head and neck. Oral Oncol. 2018 Sep;84:46-51. doi: 10.1016/j.oraloncology.2018.06.028. Epub 2018 Jul 19. PMID 30115475
- [Background] Li F, Zhang H, He M, Liao J, Chen N, Li Y, Zhou S, Palmisano M, Yu A, Pai MP, Yuan H, Sun D. Different Nanoformulations Alter the Tissue Distribution of Paclitaxel, Which Aligns with Reported Distinct Efficacy and Safety Profiles. Mol Pharm. 2018 Oct 1;15(10):4505-4516. doi: 10.1021/acs.molpharmaceut.8b00527. Epub 2018 Sep 21. PMID 30180593
- [Background] Pelzer U, Wislocka L, Juhling A, Striefler J, Klein F, Roemmler-Zehrer J, Sinn M, Denecke T, Bahra M, Riess H. Safety and efficacy of Nab-paclitaxel plus gemcitabine in patients with advanced pancreatic cancer suffering from cholestatic hyperbilirubinaemia-A retrospective analysis. Eur J Cancer. 2018 Sep;100:85-93. doi: 10.1016/j.ejca.2018.06.001. Epub 2018 Jul 4. PMID 30014884
- [Background] Metts JL, Alazraki AL, Clark D, Amankwah EK, Wasilewski-Masker KJ, George BA, Olson TA, Cash T. Gemcitabine/nab-paclitaxel for pediatric relapsed/refractory sarcomas. Pediatr Blood Cancer. 2018 Sep;65(9):e27246. doi: 10.1002/pbc.27246. Epub 2018 May 17. PMID 29770997
- [Background] Langer CJ, Kim ES, Anderson EC, Jotte RM, Modiano M, Haggstrom DE, Socoteanu MP, Smith DA, Dakhil C, Konduri K, Berry T, Ong TJ, Sanford A, Amiri K, Goldman JW, Weiss J; ABOUND.70+ Investigators. nab-Paclitaxel-Based Therapy in Underserved Patient Populations: The ABOUND.70+ Study in Elderly Patients With Advanced NSCLC. Front Oncol. 2018 Jul 24;8:262. doi: 10.3389/fonc.2018.00262. eCollection 2018. PMID 30087851
- [Background] Gajra A, Karim NA, Mulford DA, Villaruz LC, Matrana MR, Ali HY, Santos ES, Berry T, Ong TJ, Sanford A, Amiri K, Spigel DR. nab-Paclitaxel-Based Therapy in Underserved Patient Populations: The ABOUND.PS2 Study in Patients With NSCLC and a Performance Status of 2. Front Oncol. 2018 Jul 24;8:253. doi: 10.3389/fonc.2018.00253. eCollection 2018. PMID 30087850
- [Background] Cartwright TH, Parisi M, Espirito JL, Wilson TW, Pelletier C, Patel M, Babiker HM. Clinical Outcomes with First-Line Chemotherapy in a Large Retrospective Study of Patients with Metastatic Pancreatic Cancer Treated in a US Community Oncology Setting. Drugs Real World Outcomes. 2018 Sep;5(3):149-159. doi: 10.1007/s40801-018-0137-x. PMID 29946913
- [Background] Moreno L, Casanova M, Chisholm JC, Berlanga P, Chastagner PB, Baruchel S, Amoroso L, Gallego Melcon S, Gerber NU, Bisogno G, Fagioli F, Geoerger B, Glade Bender JL, Aerts I, Bergeron C, Hingorani P, Elias I, Simcock M, Ferrara S, Le Bruchec Y, Slepetis R, Chen N, Vassal G. Phase I results of a phase I/II study of weekly nab-paclitaxel in paediatric patients with recurrent/refractory solid tumours: A collaboration with innovative therapies for children with cancer. Eur J Cancer. 2018 Sep;100:27-34. doi: 10.1016/j.ejca.2018.05.002. Epub 2018 Jun 21. PMID 29936064
- [Background] Young R, Mainwaring P, Clingan P, Parnis FX, Asghari G, Beale P, Aly A, Botteman M, Romano A, Ferrara S, Margunato-Debay S, Harris M. nab-Paclitaxel plus gemcitabine in metastatic pancreatic adenocarcinoma: Australian subset analyses of the phase III MPACT trial. Asia Pac J Clin Oncol. 2018 Oct;14(5):e325-e331. doi: 10.1111/ajco.12999. Epub 2018 Jun 22. PMID 29932294
- [Background] Topcul M, Ceti N IL, Ozbas Turan S, Kolusayin Ozar MO. In vitro cytotoxic effect of PARP inhibitor alone and in combination with nab-paclitaxel on triple-negative and luminal A breast cancer cells. Oncol Rep. 2018 Jul;40(1):527-535. doi: 10.3892/or.2018.6364. Epub 2018 Apr 12. PMID 29658592
- [Background] Neumann CCM, von Horschelmann E, Reutzel-Selke A, Seidel E, Sauer IM, Pratschke J, Bahra M, Schmuck RB. Tumor-stromal cross-talk modulating the therapeutic response in pancreatic cancer. Hepatobiliary Pancreat Dis Int. 2018 Oct;17(5):461-472. doi: 10.1016/j.hbpd.2018.09.004. Epub 2018 Sep 7. PMID 30243879
- [Background] Veenstra VL, Damhofer H, Waasdorp C, van Rijssen LB, van de Vijver MJ, Dijk F, Wilmink HW, Besselink MG, Busch OR, Chang DK, Bailey PJ, Biankin AV, Kocher HM, Medema JP, Li JS, Jiang R, Pierce DW, van Laarhoven HWM, Bijlsma MF. ADAM12 is a circulating marker for stromal activation in pancreatic cancer and predicts response to chemotherapy. Oncogenesis. 2018 Nov 16;7(11):87. doi: 10.1038/s41389-018-0096-9. PMID 30442938
- [Background] Morgensztern D, Cobo M, Ponce Aix S, Postmus PE, Lewanski CR, Bennouna J, Fischer JR, Juan-Vidal O, Stewart DJ, Fasola G, Ardizzoni A, Bhore R, Wolfsteiner M, Talbot DC, Jin Ong T, Govindan R, On Behalf Of The Abound L Investigators. ABOUND.2L+: A randomized phase 2 study of nanoparticle albumin-bound paclitaxel with or without CC-486 as second-line treatment for advanced nonsquamous non-small cell lung cancer (NSCLC). Cancer. 2018 Dec 15;124(24):4667-4675. doi: 10.1002/cncr.31779. Epub 2018 Nov 1. PMID 30383906
- [Background] Marschner N, Salat C, Soling U, Hansen R, Grebhardt S, Harde J, Nusch A, Potthoff K. Final Effectiveness and Safety Results of NABUCCO: Real-World Data From a Noninterventional, Prospective, Multicenter Study in 697 Patients With Metastatic Breast Cancer Treated With nab-Paclitaxel. Clin Breast Cancer. 2018 Dec;18(6):e1323-e1337. doi: 10.1016/j.clbc.2018.07.010. Epub 2018 Aug 10. PMID 30100104
- [Background] Watson S, de la Fouchardiere C, Kim S, Cohen R, Bachet JB, Tournigand C, Ferraz JM, Lefevre M, Colin D, Svrcek M, Meurisse A, Louvet C. Oxaliplatin, 5-Fluorouracil and Nab-paclitaxel as perioperative regimen in patients with resectable gastric adenocarcinoma: A GERCOR phase II study (FOXAGAST). Eur J Cancer. 2019 Jan;107:46-52. doi: 10.1016/j.ejca.2018.11.006. Epub 2018 Dec 7. PMID 30529902
- [Background] Li YF, Zhang C, Zhou S, He M, Zhang H, Chen N, Li F, Luan X, Pai M, Yuan H, Sun D, Li Y. Species difference in paclitaxel disposition correlated with poor pharmacological efficacy translation from mice to humans. Clin Pharmacol. 2018 Nov 8;10:165-174. doi: 10.2147/CPAA.S185449. eCollection 2018. PMID 30519122
- [Background] Hurria A, Soto-Perez-de-Celis E, Blanchard S, Burhenn P, Yeon CH, Yuan Y, Li D, Katheria V, Waisman JR, Luu TH, Somlo G, Noonan AM, Lee T, Sudan N, Chung S, Rotter A, Arsenyan A, Levi A, Choi J, Rubalcava A, Morrison R, Mortimer JE. A Phase II Trial of Older Adults With Metastatic Breast Cancer Receiving nab-Paclitaxel: Melding the Fields of Geriatrics and Oncology. Clin Breast Cancer. 2019 Apr;19(2):89-96. doi: 10.1016/j.clbc.2018.10.002. Epub 2018 Oct 16. PMID 30503309
- [Background] Fernandez A, Salgado M, Garcia A, Buxo E, Vera R, Adeva J, Jimenez-Fonseca P, Quintero G, Llorca C, Canabate M, Lopez LJ, Munoz A, Ramirez P, Gonzalez P, Lopez C, Reboredo M, Gallardo E, Sanchez-Canovas M, Gallego J, Guillen C, Ruiz-Miravet N, Navarro-Perez V, De la Camara J, Ales-Diaz I, Pazo-Cid RA, Carmona-Bayonas A. Prognostic factors for survival with nab-paclitaxel plus gemcitabine in metastatic pancreatic cancer in real-life practice: the ANICE-PaC study. BMC Cancer. 2018 Nov 29;18(1):1185. doi: 10.1186/s12885-018-5101-3. PMID 30497432
- [Background] Awasthi N, Schwarz MA, Zhang C, Schwarz RE. Augmentation of Nab-Paclitaxel Chemotherapy Response by Mechanistically Diverse Antiangiogenic Agents in Preclinical Gastric Cancer Models. Mol Cancer Ther. 2018 Nov;17(11):2353-2364. doi: 10.1158/1535-7163.MCT-18-0489. Epub 2018 Aug 30. PMID 30166402
- [Background] Nakao A, Uchino J, Igata F, On R, Ikeda T, Yatsugi H, Hirano R, Sasaki T, Tanimura K, Imabayashi T, Tamiya N, Kaneko Y, Yamada T, Nagata N, Watanabe K, Kishimoto J, Takayama K, Fujita M. Nab-paclitaxel maintenance therapy following carboplatin + nab-paclitaxel combination therapy in chemotherapy naive patients with advanced non-small cell lung cancer: multicenter, open-label, single-arm phase II trial. Invest New Drugs. 2018 Oct;36(5):903-910. doi: 10.1007/s10637-018-0617-6. Epub 2018 May 30. PMID 29846848
- [Background] Cristea MC, Frankel P, Synold T, Rivkin S, Lim D, Chung V, Chao J, Wakabayashi M, Paz B, Han E, Lin P, Leong L, Hakim A, Carroll M, Prakash N, Dellinger T, Park M, Morgan RJ. A phase I trial of intraperitoneal nab-paclitaxel in the treatment of advanced malignancies primarily confined to the peritoneal cavity. Cancer Chemother Pharmacol. 2019 Mar;83(3):589-598. doi: 10.1007/s00280-019-03767-9. Epub 2019 Jan 8. PMID 30623229
- [Background] Hegewisch-Becker S, Aldaoud A, Wolf T, Krammer-Steiner B, Linde H, Scheiner-Sparna R, Hamm D, Janicke M, Marschner N; TPK-Group (Tumour Registry Pancreatic Cancer). Results from the prospective German TPK clinical cohort study: Treatment algorithms and survival of 1,174 patients with locally advanced, inoperable, or metastatic pancreatic ductal adenocarcinoma. Int J Cancer. 2019 Mar 1;144(5):981-990. doi: 10.1002/ijc.31751. Epub 2018 Oct 3. PMID 30006989
- [Background] Wang Z, Huang C, Yang JJ, Song Y, Cheng Y, Chen GY, Yan HH, Ben XS, Wang BC, Xu CR, Jiang BY, Zhou Q, Chen HJ, Wu YL. A randomised phase II clinical trial of nab-paclitaxel and carboplatin compared with gemcitabine and carboplatin as first-line therapy in advanced squamous cell lung carcinoma (C-TONG1002). Eur J Cancer. 2019 Mar;109:183-191. doi: 10.1016/j.ejca.2019.01.007. Epub 2019 Feb 7. PMID 30739019
- [Background] Woo W, Carey ET, Choi M. Spotlight on liposomal irinotecan for metastatic pancreatic cancer: patient selection and perspectives. Onco Targets Ther. 2019 Feb 21;12:1455-1463. doi: 10.2147/OTT.S167590. eCollection 2019. PMID 30863113
- [Background] Seiwert TY, Foster CC, Blair EA, Karrison TG, Agrawal N, Melotek JM, Portugal L, Brisson RJ, Dekker A, Kochanny S, Gooi Z, Lingen MW, Villaflor VM, Ginat DT, Haraf DJ, Vokes EE. OPTIMA: a phase II dose and volume de-escalation trial for human papillomavirus-positive oropharyngeal cancer. Ann Oncol. 2019 Feb 1;30(2):297-302. doi: 10.1093/annonc/mdy522. PMID 30481287
- [Background] De Luca R, Profita G, Cicero G. Nab-paclitaxel in pretreated metastatic breast cancer: evaluation of activity, safety, and quality of life. Onco Targets Ther. 2019 Feb 26;12:1621-1627. doi: 10.2147/OTT.S191519. eCollection 2019. PMID 30881017
- [Background] Morgensztern D, Ko A, O'Brien M, Ong TJ, Waqar SN, Socinski MA, Postmus PE, Bhore R. Association between depth of response and survival in patients with advanced-stage non-small cell lung cancer treated with first-line chemotherapy. Cancer. 2019 Jul 15;125(14):2394-2399. doi: 10.1002/cncr.32114. Epub 2019 Apr 1. PMID 30933354
- [Background] Li F, Yuan H, Zhang H, He M, Liao J, Chen N, Li Y, Zhou S, Palmisano M, Yu A, Pai M, Sun D. Neonatal Fc Receptor (FcRn) Enhances Tissue Distribution and Prevents Excretion of nab-Paclitaxel. Mol Pharm. 2019 Jun 3;16(6):2385-2393. doi: 10.1021/acs.molpharmaceut.8b01314. Epub 2019 May 1. PMID 31002261
- [Background] Sonbol MB, Ahn DH, Goldstein D, Okusaka T, Tabernero J, Macarulla T, Reni M, Li CP, O'Neil B, Van Cutsem E, Bekaii-Saab T. CanStem111P trial: a Phase III study of napabucasin plus nab-paclitaxel with gemcitabine. Future Oncol. 2019 Apr;15(12):1295-1302. doi: 10.2217/fon-2018-0903. Epub 2019 Feb 15. PMID 30768369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 87 sites in Germany, Italy, Spain, the United Kingdom and the United States.
Pre-assignment Details: Participants with a response or stable disease during Induction were randomised 2:1 into investigative treatment (nab-paclitaxel plus best supportive care [BSC] or BSC only) stratified by disease stage, response during induction and Eastern Cooperative Oncology Group (ECOG) performance status.
Groups:
- All Participants - Induction: During induction, participants received nab-paclitaxel plus carboplatin as standard of care: nab-paclitaxel 100 mg/m^2 IV infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle and carboplatin AUC = 6 mg*min/mL IV on Day 1 of each 21-day cycle. If the participant had radiological or clinical progressive disease (PD), they were discontinued from the study and not followed. If the participant had a complete response, partial response, or stable disease without PD at the end of 4 cycles, he/she were eligible to be randomised to the maintenance phase
- Nab-Paclitaxel + Best Supportive Care (BSC): Maintenance Phase: Following randomization, participants in this treatment arm were administered nab-paclitaxel 100 mg/m^2 by IV infusion over 30 minutes on Days 1 and 8 of each 21-day cycle, plus best supportive care until disease progression.
- Best Supportive Care (BSC): Maintenance Phase: Following randomization, participants in this treatment arm were administered best supportive care (only) until disease progression.
Period: Induction
Arm/Group | All Participants - Induction | Nab-Paclitaxel + Best Supportive Care (BSC) | Best Supportive Care (BSC)
Started | 427 | 0 | 0
Received Study Drug | 420 | 0 | 0
Completed (Completed = participants who continued to maintenance period.) | 202 (If radiologically CR, PR or SD after 4 cycles of treatment, participants continue on to Maintenance.) | 0 | 0
Not Completed | 225 | 0 | 0
Not completed — Never treated | 7 | 0 | 0
Not completed — Progressive disease | 77 | 0 | 0
Not completed — Adverse Event | 51 | 0 | 0
Not completed — Withdrawal by Subject | 22 | 0 | 0
Not completed — Death | 21 | 0 | 0
Not completed — Symptomatic deterioration | 16 | 0 | 0
Not completed — Study terminated by sponsor | 12 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Miscellaneous | 14 | 0 | 0
Not completed — Induction Treatment Ongoing | 4 | 0 | 0
Period: Maintenance
Arm/Group | All Participants - Induction | Nab-Paclitaxel + Best Supportive Care (BSC) | Best Supportive Care (BSC)
Started | 0 | 136 | 66
Completed (Completed = Participants who continued on treatment) | 0 | 12 | 6
Not Completed | 0 | 124 | 60
Not completed — Death | 0 | 3 | 2
Not completed — Adverse Event | 0 | 21 | 1
Not completed — Progressive disease | 0 | 84 | 47
Not completed — Symptomatic deterioration | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 5
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Other | 0 | 6 | 3
Period: Survival Follow-up
Arm/Group | All Participants - Induction | Nab-Paclitaxel + Best Supportive Care (BSC) | Best Supportive Care (BSC)
Started | 0 | 117 (Participants are not taking study intervention but are on appropriate standard of care.) | 55 (Participants are not taking study intervention but are on appropriate standard of care.)
Completed (Completed = Participants alive to end of study) | 0 | 38 | 9
Not Completed | 0 | 79 | 46
Not completed — Death | 0 | 78 | 45
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Induction includes participants who were enrolled and treated however, baseline characteristics (BLC) for non-randomised participants is not displayed. The total number represents the ITT population in the maintenance phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nab-Paclitaxel + Best Supportive Care (BSC) | Best Supportive Care (BSC) | Total
Number analyzed (Participants) | 136 | 66 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] — Continuous age values in Total column represent the 202 participants in the Maintenance Period. Induction includes participants who were enrolled and treated however, baseline characteristics for non-randomised participants is not displayed. The total number represents the ITT population in the maintenance phase.
  years | 67.1 (9.02) | 66.8 (8.06) | 67.0 (8.70)
Age, Customized [Count of Participants; unit: Participants] — Induction includes participants who were enrolled and treated in the induction phase. Baseline characteristics are displayed only for participants randomised in the maintenance phase. The total number represents the ITT population in the maintenance phase.
  Participants
    <65 years | 48 | 27 | 75
    >=65 years | 88 | 39 | 127
    <70 years | 79 | 41 | 120
    >=70 years | 57 | 25 | 82
    <75 years | 110 | 55 | 165
    >=75 years | 26 | 11 | 37
Sex: Female, Male [Count of Participants; unit: Participants] — Induction includes participants who were enrolled and treated in the induction phase. Baseline characteristics are displayed only for participants randomised in the maintenance phase. The total number represents the ITT population in the maintenance phase.
  Participants
    Female | 49 | 23 | 72
    Male | 87 | 43 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Induction includes participants who were enrolled and treated in the induction phase. Baseline characteristics are displayed only for participants randomized in the maintenance phase. The total number represents the ITT population in the maintenance phase.
  Participants
    Hispanic or Latino | 3 | 5 | 8
    Not Hispanic or Latino | 132 | 61 | 193
    Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Induction includes participants who were enrolled and treated in the induction phase. Baseline characteristics are displayed only for participants randomized in the maintenance phase. The total number represents the ITT population in the maintenance phase.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Black or African American | 9 | 2 | 11
    White | 125 | 62 | 187
    Other | 0 | 2 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG PS assesses how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. - 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled. Baseline characteristics are displayed only for participants randomized in the maintenance phase. The total number represents the ITT population in the maintenance phase.
  Participants
    0=fully active, no restriction | 41 | 19 | 60
    1=fully ambulatory; restricted strenuous activity | 95 | 47 | 142
    >=2=ambulatory/self care; no work or worse | 0 | 0 | 0
Overall Tumor Response at End of Induction [Count of Participants; unit: Participants] — Tumor response to Induction part chemotherapy for stratification is the response assessed at the last computed tomography (CT) scan before randomization. Baseline characteristics are displayed only for participants randomized in the maintenance phase. The total number represents the ITT population in the maintenance phase.
  Participants
    Complete response | 1 | 2 | 3
    Partial response | 92 | 42 | 134
    Stable disease | 41 | 21 | 62
    Progressive disease | 2 | 0 | 2
    Not evaluable | 0 | 1 | 1
Confirmed Histology [Count of Participants; unit: Participants] — The histology categories included those with a tumor histology of squamous versus non-squamous types. Baseline characteristics for non-randomized participants is not displayed. The total number represents the ITT population in the maintenance phase.
  Participants
    Squamous cell carcinoma | 136 | 66 | 202
    Squamous cell carcinoma not confirmed | 0 | 0 | 0
Disease Stage at Enrollment [Count of Participants; unit: Participants] — Disease stage = how big the tumor is and how far it has spread. Disease stages range from 0 (not spread) to IV (spread throughout the body). Stage 0: the cancer has not spread beyond the inner lining of the lung. Stage I: the cancer is small and hasn't spread to the lymph nodes (LN). Stage II: the cancer has spread to some LN near the original tumor. Stage III: the cancer has spread to nearby tissue or spread to far away LN. Stage IV: the cancer has spread to other organs such as lung, brain, or liver. BLC are displayed for participants randomized in the maintenance phase.
  Participants
    Stage IIIB | 18 | 8 | 26
    Stage IV | 118 | 58 | 176

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS) From Randomization Into Maintenance
Description: Progression-free survival is defined as the time in months from the date of randomization to the date of disease progression based on the investigator's assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria (documented by computerized axial tomography [CT scan], not including symptomatic deterioration) or death (any cause) on or prior to 01 Aug 2019. RECIST 1.1 Definition: - Complete response (CR) -disappearance of all target lesions; - Partial response (PR) -at least a 30% decrease in the sum of diameters of target lesions from baseline - Stable disease (SD) -neither sufficient shrinkage to qualify for partial response (PR) nor sufficient increase of lesions to qualify for progressive disease (PD) - Progressive Disease (PD) - At least a 20% increase in the sum of diameters of target lesions from nadir, and/or the appearance of new lesions.
Time Frame: From the date of randomization to the date of disease progression or death of any cause; up to data cut off date of 15 September 2017; up to 27.6 months
Population: Intent to treat (ITT) population of participants randomized to Maintenance. The ITT population in the Maintenance part included all randomized subjects regardless of whether the subject received any study drug or had any efficacy assessments collected.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel + Best Supportive Care (BSC) | Best Supportive Care (BSC)
Number analyzed (Participants) | 136 | 66
months | 3.12 [2.73 to 4.60] | 2.60 [1.64 to 3.45]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + Best Supportive Care (BSC) vs Best Supportive Care (BSC); 5% level of significance. Hazard ratio is based on stratified Cox proportional hazards regression model. The following stratification factors were evaluated in the sparse strata elimination algorithm: stage of disease (IIIB or IV) at diagnosis, ECOG performance status (0 or 1) at end of Induction, and tumor response (CR/PR or SD) at the end of Induction; Test type: Superiority; p = 0.3486, stratified log-rank test — Stratification factors evaluated in the sparse strata elimination algorithm: stage of disease (IIIB or IV) at diagnosis, ECOG performance status (0 or 1) at end of Induction, and tumor response (CR/PR or SD) at end of Induction; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.61 to 1.19] — Hazard ratio: nab-paclitaxel + BSC / BSC Alone

2. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS) From Randomization Into Maintenance
Description: Overall survival was defined as the duration in months between randomization and death from any cause. Participants who were still alive as of the clinical cut-off date had their OS censored at the date of last contact or clinical cut-off (01 August 2019 whichever was earlier. The last contact date was the date of the last record in the database, or if the subject was lost to follow-up, the last known date that the subject was alive.
Time Frame: From the date of randomization to death from any cause; up to 01 August 2019; survival follow up was 55.89 months
Population: Intent to Treat population of participants randomized to maintenance.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel + Best Supportive Care (BSC) | Best Supportive Care (BSC)
Number analyzed (Participants) | 136 | 66
months | 17.61 [13.86 to 21.09] | 12.16 [7.56 to 18.99]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + Best Supportive Care (BSC) vs Best Supportive Care (BSC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0365, stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.47 to 0.98] — Hazard ratio: nab-paclitaxel + BSC / BSC Alone

3. Secondary Outcome: Percentage of Participants Who Achieved a Confirmed Overall Response of Complete Response or Partial Response (Overall Response Rate) Over Entire Study
Description: Overall response was defined as the percentage of participants with a confirmed assessment of complete response (CR) or partial response (PR) according to RECIST 1.1 criteria and confirmed in no less than 28 days. The 95% confidence interval (CI) was calculated using Clopper-Pearson method. RECIST 1.1 Definition: - Complete response-disappearance of all target lesions; any pathological lymph nodes (whether target or non target) must have reduction in short axis to < 10 mm. - Partial response-at least a 30% decrease in the sum of diameters of target lesions from baseline.
Time Frame: Day 1 of treatment in the induction period and subsequent anticancer therapy, death or discontinuation up to 01 August 2019; maximum treatment duration was 234.1 weeks for entire study
Population: Intent to treat population of participants randomized to Maintenance
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Nab-Paclitaxel + BSC: Induction + Maintenance: Participants randomized to this treatment arm for Maintenance, inclusive of their experience during Induction. During induction, participants received nab-paclitaxel plus carboplatin as standard of care: nab-paclitaxel 100 mg/m^2 IV infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle and carboplatin AUC = 6 mg*min/mL IV on Day 1 of each 21-day cycle. If the participant had a complete response, partial response, or stable disease without PD at the end of 4 cycles, he/she continued to the maintenance phase. Maintenance: Following randomization, participants in this treatment arm were administered nab-paclitaxel 100 mg/m^2 by IV infusion over 30 minutes on Days 1 and 8 of each 21-day cycle, plus best supportive care until disease progression.
- BSC: Induction + Maintenance: Participants randomized to this treatment arm for Maintenance, inclusive of their experience during Induction. During induction, participants received nab-paclitaxel plus carboplatin as standard of care: nab-paclitaxel 100 mg/m^2 IV infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle and carboplatin AUC = 6 mg*min/mL IV on Day 1 of each 21-day cycle. If the participant had a complete response, partial response, or stable disease without PD at the end of 4 cycles, he/she continued to the maintenance phase. Maintenance: Following randomization, participants in this treatment arm were administered best supportive care (only) until disease progression.
Arm/Group | Nab-Paclitaxel + BSC: Induction + Maintenance | BSC: Induction + Maintenance
Number analyzed (Participants) | 136 | 66
percentage of participants | 69.1 [60.6 to 76.8] | 57.6 [44.8 to 69.7]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + BSC: Induction + Maintenance vs BSC: Induction + Maintenance; 5% level of significance. The rate ratio and its 95% CI were based on the non-stratified analysis; Test type: Superiority; p = 0.0870, Cochran-Mantel-Haenszel — Stratification factors evaluated in the sparse strata elimination algorithm: stage of disease (IIIB or IV) at diagnosis, ECOG performance status (0 or 1) at the end of Induction, and tumor response (CR/PR or SD) at the end of Induction; Overall response rate ratio = 1.20, 95% CI 2-sided [0.948 to 1.519] — response ratio: nab-paclitaxel + BSC / BSC Alone

4. Secondary Outcome: Kaplan-Meier Estimate of Progression-Free Survival (PFS) Over Entire Study
Description: PFS was defined as the time in months from Day 1 of treatment for the Induction part to the date of disease progression according to RECIST 1.1 criteria (documented by CT-scan, not including symptomatic deterioration) or death (any cause) on or prior to 01 August 2019, whichever occurred earlier. RECIST 1.1 Definition: - Progressive Disease (PD) - At least a 20% increase in the sum of diameters of target lesions from nadir; the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of new lesions is also considered progression.
Time Frame: Between Day 1 of the Induction Part through to the date of disease progression or death; up to 01 August 2019; the maximum treatment duration was 234.1 weeks for entire study
Population: Intent to treat population of participants randomized to Maintenance
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel + BSC: Induction + Maintenance | BSC: Induction + Maintenance
Number analyzed (Participants) | 136 | 66
months | 6.47 [5.65 to 7.79] | 5.55 [4.96 to 6.67]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + BSC: Induction + Maintenance vs BSC: Induction + Maintenance; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4164, stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.62 to 1.22] — Hazard ratio: nab-paclitaxel + BSC / BSC Alone

5. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS) Over Entire Study
Description: Overall survival was defined as the time in months from Day 1 of treatment for the Induction part to death from any cause. Subjects who were alive at the time of analysis had their OS censored at the date or last contact of 01 August 2019, whichever was earlier. The last contact date was the date of the last record in the database, or if the subject was lost to follow-up, the last known date that the subject was alive.
Time Frame: Between Day 1 of treatment in the Induction Part to death from any cause; up to 01 August 2019; survival follow up was 55.89 months
Population: ITT population of participants randomized to Maintenance.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel + BSC: Induction + Maintenance | BSC: Induction + Maintenance
Number analyzed (Participants) | 136 | 66
months | 20.57 [17.05 to 24.05] | 15.05 [10.81 to 22.14]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + BSC: Induction + Maintenance vs BSC: Induction + Maintenance; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0381, stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.47 to 0.98] — Hazard ratio: nab-paclitaxel + BSC / BSC Alone

6. Secondary Outcome: Percentage of Participants Who Achieved a Confirmed Overall Response of Complete Response or Partial Response (Overall Response Rate) In Maintenance Beyond the Response in Induction
Description: Overall response in the maintenance period was defined as the percentage of participants who showed an improvement in best overall response from stable disease (SD) or partial response (PR) during Induction to a Complete Response (CR) or PR during Maintenance according to RECIST 1.1 criteria and confirmed in no less than 28 days. Evaluation takes as reference the lesion measurement or status at the last tumor assessment before randomization to Maintenance. The 95% CI was calculated using Clopper-Pearson method. RECIST 1.1 Definition: - Complete response-disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. - Partial response-at least a 30% decrease in the sum of diameters of target lesions from baseline. - Stable disease-neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease.
Time Frame: For the induction period the maximum treatment was 19 weeks for the maintenance period the maximum treatment was 150 weeks.
Population: Intent to treat population of participants randomized to the maintenance period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nab-Paclitaxel + BSC: Induction + Maintenance | BSC: Induction + Maintenance
Number analyzed (Participants) | 136 | 66
percentage of participants | 9.6 [5.2 to 15.8] | 3.0 [0.4 to 10.5]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + BSC: Induction + Maintenance vs BSC: Induction + Maintenance; Test type: Superiority; p = 0.0978, Cochran-Mantel-Haenszel — 5% level of significance; Overall response rate ratio = 3.15, 95% CI 2-sided [0.733 to 13.574] — Response rate ratio: nab-paclitaxel + BSC / BSC Alone

7. Secondary Outcome: Percentage of Participants Who Achieved Disease Control (Disease Control Rate) by Investigator Assessment During Induction and Over the Entire Study
Description: Disease control rate was defined as the percentage of participants who had radiologic CR, PR or SD for >= 6 weeks according to RECIST 1.1 criteria as determined by the investigator. Only participants with a confirmed CR/PR are included in this summary. Two timeframes are offered: - Time to confirmed response within the Induction timeframe. - Time to Confirmed Response Over the Entire Study, i.e. the time from Day 1 of treatment in Induction to the first occurrence of confirmed CR/PR any time during the study. RECIST 1.1 Definition: - CR- disappearance of all target lesions; any pathological lymph nodes (whether target or non target) must have reduction in short axis to < 10 mm. - PR- at least a 30% decrease in the sum of diameters of target lesions from baseline; - SD- neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for PD. The 95% CI was calculated using Clopper-Pearson method.
Time Frame: Induction is from Day 1 to a maximum treatment time of 19 weeks; entire study from Day 1 induction through maintenance up to PD; up to 01 August 2019; maximum treatment duration was 234.1 weeks for entire study
Population: Induction includes the ITT population of participants treated during Induction. Entire Study includes the entire experience of the ITT population of participants randomized to maintenance.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Nab-Paclitaxel + BSC: Induction + Maintenance: Participants randomized to this treatment arm for Maintenance, inclusive of their experience during Induction. During induction, During induction, participants received nab-paclitaxel plus carboplatin as standard of care: nab-paclitaxel 100 mg/m^2 IV infusion over 30 minutes on Days 1, 8, and 15 of each 21-day cycle and carboplatin AUC = 6 mg*min/mL IV on Day 1 of each 21-day cycle. If the participant had a complete response, partial response, or stable disease without PD at the end of 4 cycles, he/she continued to the maintenance phase. Maintenance: Following randomization, participants in this treatment arm were administered nab-paclitaxel 100 mg/m^2 by IV infusion over 30 minutes on Days 1 and 8 of each 21-day cycle, plus best supportive care until disease progression.
Arm/Group | All Participants - Induction | Nab-Paclitaxel + BSC: Induction + Maintenance | BSC: Induction + Maintenance
Number analyzed (Participants) | 420 | 136 | 66
percentage of participants | 47.9 [43.0 to 52.8] | 99.3 [96.0 to 100.0] | 100.0 [94.6 to 100.0]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + BSC: Induction + Maintenance vs BSC: Induction + Maintenance; The rate ratio and its 95% confidence interval are based on non-stratified analysis; Test type: Superiority; disease control rate ratio = 0.99, 95% CI 2-sided [0.978 to 1.007] — Disease control rate ratio: nab-paclitaxel + BSC / BSC Alone

8. Secondary Outcome: Time to Confirmed Response During Induction and Over the Entire Study
Description: Time to confirmed complete or partial response (CR/PR) is defined as the time from day 1 of treatment in Induction to the first occurrence of confirmed CR/PR. Two timeframes are offered: - Time to confirmed response within the Induction timeframe. - Time to Confirmed Response Over the Entire Study, i.e. the time from Day 1 of treatment in Induction to the first occurrence of confirmed CR/PR any time during the study. Only participants with a confirmed CR or PR are included in this summary.
Time Frame: as for outcome 7
Population: Includes the ITT population of participants who had a response. Induction includes the ITT population of participants treated during Induction who had a response. Induction+Maintenance includes the ITT population of participants randomized to Maintenance who had a response.
Measure: Median (Full Range); unit: months
Arm/Group | All Participants - Induction | Nab-Paclitaxel + BSC: Induction + Maintenance | BSC: Induction + Maintenance
Number analyzed (Participants) | 126 | 94 | 38
months | 1.446 [1.15 to 4.60] | 1.478 [1.15 to 8.51] | 1.413 [1.18 to 4.21]

9. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response Over the Entire Study
Description: Duration of overall response was measured from the time criteria were first met for CR/PR until the first date the recurrent or progressive disease (PD) was radiologically documented. Participants who did not have PD after the response were censored on the date of last tumor assessment. If a participant died before PD, the participant was censored on the date of death.
Time Frame: Between Day 1 of the Induction Period through to the date of disease progression or death; up to 01 August 2019; maximum treatment duration was 234.1 weeks for entire study.
Population: The ITT population of participants randomized to the maintenance period and had a confirmed partial or complete response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-Paclitaxel + BSC: Induction + Maintenance | BSC: Induction + Maintenance
Number analyzed (Participants) | 94 | 38
months | 5.95 [4.60 to 7.06] | 4.60 [3.68 to 5.49]
Statistical Analysis 1: Comparison: Nab-Paclitaxel + BSC: Induction + Maintenance vs BSC: Induction + Maintenance; Hazard ratio was based on stratified Cox proportional hazards regression model. The following stratification factors were evaluated in the sparse strata elimination algorithm: stage of disease (IIIB or IV) at diagnosis, ECOG performance status (0 or 1) at the end of Induction, and tumor response (CR/PR or SD) at the end of Induction; Test type: Superiority; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.59 to 1.47] — Hazard ratio: nab-paclitaxel + BSC / BSC Alone

10. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs) in the Induction Period
Description: TEAE in the Induction part is defined as any adverse event (AE) with an onset on or after Day 1 of treatment for the Induction part, and on or before the day of randomization for subjects who entered into the Maintenance part, or, for subjects who did not enter into the Maintenance part, before the treatment discontinuation date plus 28 days or any serious AE which occurred thereafter but was determined to be related to any study drug by the investigator. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and the scale: Grade 1 = Mild, Grade 2 = Moderate Grade, 3 = Severe Grade, 4 = Life threatening, Grade 5 = Death. Relation to study drug was determined by the investigator.
Time Frame: Day 1 of Induction up to Week 23 (maximum treatment in Induction plus 4 weeks if not continuing into Maintenance)
Population: Safety population of participants treated during induction period.
Measure: Count of Participants; unit: Participants
Groups:
- TEAE Specific to Nab-Paclitaxel: TEAE categories specific to nab-paclitaxel intervention as determined by the investigator.
- TEAE Specific to Carboplatin: TEAE categories specific to carboplatin intervention as determined by the investigator.
Arm/Group | All Participants - Induction | TEAE Specific to Nab-Paclitaxel | TEAE Specific to Carboplatin
Number analyzed (Participants) | 420 | 420 | 420
Participants
  TEAE | 419 | NA — category not specific to study intervention | NA — category not specific to study intervention
  Serious TEAE | 177 | NA — category not specific to study intervention | NA — category not specific to study intervention
  Severity Grade 3/4 TEAE | 337 | NA — category not specific to study intervention | NA — category not specific to study intervention
  Severity Grade 3 or higher TEAE | 340 | NA — category not specific to study intervention | NA — category not specific to study intervention
  Treatment-related (trt-related) TEAE | 408 | 407 | 394
  Trt-related serious TEAE | 82 | 80 | 73
  TEAE-study drug dose reduced or interrupted | 341 | 340 | 291
  Trt-related TEAE-dose reduced or interrupted | 301 | 292 | 236
  TEAE-study drug withdrawn | 55 | 55 | 53
  Trt-related TEAE-study drug withdrawn | 35 | 34 | 29
  TEAE-outcome of death | 32 | NA — category not specific to study intervention | NA — category not specific to study intervention
  Trt-related TEAE-outcome of death | 7 | 7 | 6

11. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs) Over the Entire Study
Description: TEAE over entire study is defined as any adverse event (AE) with an onset on or after Day 1 of treatment for the Induction part, and before the treatment discontinuation date plus 28 days, or any serious AE which occurred thereafter but was determined to be related to any study drug by the investigator. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and the scale: Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life threatening, Grade 5 = Death. Relation to study drug was determined by the investigator.
Time Frame: From Day 1 up to 01 August 2019; (maximum treatment length plus 28 days); the maximum treatment duration was 234.1 weeks for entire study
Population: Safety population of participants randomized into maintenance, inclusive of both the induction and maintenance periods.
Measure: Count of Participants; unit: Participants
Groups:
- Nab-Paclitaxel + BSC: Induction + Maintenance: Participants randomized to this treatment arm for Maintenance, inclusive of their experience during Induction. During induction, participants received nab-paclitaxel plus carboplatin as standard of care. If the participant had a complete response, partial response, or stable disease without PD at the end of 4 cycles, he/she continued to the maintenance phase. Maintenance: Following randomization, participants in this treatment arm were administered nab-paclitaxel 100 mg/m^2 by IV infusion over 30 minutes on Days 1 and 8 of each 21-day cycle, plus best supportive care until disease progression.
- Nab-Paclitaxel + BSC: TEAE Specific to Nab-Paclitaxel: TEAE categories specific to nab-paclitaxel intervention, as determined by the investigator, for participants randomized to the Nab-Paclitaxel + BSC treatment arm. Nab-paclitaxel was administered during Induction and Maintenance.
- Nab-Paclitaxel + BSC: TEAE Specific to Carboplatin: TEAE categories specific to carboplatin intervention as determined by the investigator, for participants randomized to the Nab-Paclitaxel + BSC treatment arm. Carboplatin was administered during Induction.
- Nab-Paclitaxel + BSC: TEAE Specific to BSC: TEAE categories specific to best supportive care (BSC) as determined by the investigator, for participants randomized to the Nab-Paclitaxel + BSC treatment arm. BSC was administered during Maintenance.
- BSC: Induction + Maintenance: Participants randomized to this treatment arm for Maintenance, inclusive of their experience during Induction. During induction, participants received nab-paclitaxel plus carboplatin as standard of care. If the participant had a complete response, partial response, or stable disease without PD at the end of 4 cycles, he/she continued to the maintenance phase. Maintenance: Following randomization, participants in this treatment arm were administered best supportive care (only) until disease progression.
- BSC: TEAE Specific to Nab-Paclitaxel: TEAE categories specific to nab-paclitaxel intervention, as determined by the investigator, for participants randomized to the BSC treatment arm. Nab-paclitaxel was administered during Induction.
- BSC: TEAE Specific to Carboplatin: TEAE categories specific to carboplatin intervention as determined by the investigator, for participants randomized to the BSC treatment arm. Carboplatin was administered during Induction.
- BSC: TEAE Specific to BSC: TEAE categories specific to best supportive care (BSC) as determined by the investigator, for participants randomized to the BSC treatment arm. BSC was administered during Maintenance.
Arm/Group | Nab-Paclitaxel + BSC: Induction + Maintenance | Nab-Paclitaxel + BSC: TEAE Specific to Nab-Paclitaxel | Nab-Paclitaxel + BSC: TEAE Specific to Carboplatin | Nab-Paclitaxel + BSC: TEAE Specific to BSC | BSC: Induction + Maintenance | BSC: TEAE Specific to Nab-Paclitaxel | BSC: TEAE Specific to Carboplatin | BSC: TEAE Specific to BSC
Number analyzed (Participants) | 130 | 130 | 130 | 130 | 62 | 62 | 62 | 62
Participants
  TEAE | 130 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention | 62 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention
  Serious TEAE | 54 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention | 21 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention
  Severity Grade 3/4 TEAE | 108 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention | 48 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention
  Severity Grade 3 or higher TEAE | 109 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention | 48 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention
  Treatment-related (trt-related) TEAE | 129 | 129 | 123 | 18 | 61 | 61 | 58 | 1
  Trt-related serious TEAE | 22 | 22 | 16 | 1 | 8 | 8 | 7 | 0
  TEAE-study drug dose reduced or interrupted | 115 | 113 | 95 | 17 | 52 | 52 | 45 | 1
  Trt-related TEAE-dose reduced or interrupted | 107 | 104 | 85 | 0 | 45 | 45 | 37 | 0
  TEAE-study drug withdrawn | 22 | 22 | 1 | 20 | 0 | 1 | 1 | 0
  Trt-related TEAE- study drug withdrawn | 18 | 18 | 1 | 2 | 1 | 0 | 0 | 0
  TEAE-outcome of death | 4 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention | 2 | NA — category not specific to study intervention | NA — category not specific to study intervention | NA — category not specific to study intervention
  Trt-related TEAE-outcome of death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1. All Participants - Induction: Day 1 up to 23 weeks (maximum treatment in Induction plus 4 weeks if not continuing into Maintenance) 2. Nab-Paclitaxel + Best Supportive Care (BSC): Randomization into Maintenance up to 154 weeks (maximum treatment in Maintenance plus 4 weeks) 3. Best Supportive Care (BSC): Randomization into Maintenance up to 120 weeks (maximum treatment in Maintenance plus 4 weeks) TEAEs are reported up to the data cut off date of 01 August 2019.
Description: All-Cause Mortality events are reported from the ITT population (participants who received at least 1 dose of study treatment regardless of whether they had efficacy assessments collected); up to date of 01 August 2019.
Groups:
- Nab-Paclitaxel + Best Supportive Care (Maintenance): Maintenance Phase: Following randomization, participants in this treatment arm were administered nab-paclitaxel 100 mg/m^2 by IV infusion over 30 minutes on Days 1 and 8 of each 21-day cycle, plus best supportive care until disease progression.
- Best Supportive Care (Maintenance): Maintenance Phase: Following randomization, participants in this treatment arm were administered best supportive care (only) until disease progression.
Arm/Group | All Participants - Induction | Nab-Paclitaxel + Best Supportive Care (Maintenance) | Best Supportive Care (Maintenance)
All-Cause Mortality (participants affected / at risk) | 80/420 | 82/130 | 48/62
Serious Adverse Events (participants affected / at risk) | 177/420 | 32/130 | 13/62
Other Adverse Events (participants affected / at risk) | 417/420 | 122/130 | 45/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants - Induction (N=420) | Nab-Paclitaxel + Best Supportive Care (Maintenance) (N=130) | Best Supportive Care (Maintenance) (N=62)
Anaemia (Blood and lymphatic system disorders) | 17 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 0 | 1
Atrial flutter (Cardiac disorders) | 3 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Asthenia (General disorders) | 6 | 3 | 0
Catheter site pain (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Death (General disorders) | 5 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 4 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 6 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 2 | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 4 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 3 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Paraspinal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 24 | 4 | 3
Sepsis (Infections and infestations) | 9 | 3 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspiration bronchial (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 14 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 2 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 4 | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 11 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants - Induction (N=420) | Nab-Paclitaxel + Best Supportive Care (Maintenance) (N=130) | Best Supportive Care (Maintenance) (N=62)
Anaemia (Blood and lymphatic system disorders) | 256 | 24 | 6
Leukopenia (Blood and lymphatic system disorders) | 80 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 225 | 14 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 163 | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 27 | 4 | 2
Constipation (Gastrointestinal disorders) | 130 | 14 | 0
Diarrhoea (Gastrointestinal disorders) | 158 | 18 | 4
Dyspepsia (Gastrointestinal disorders) | 37 | 3 | 1
Nausea (Gastrointestinal disorders) | 191 | 16 | 2
Stomatitis (Gastrointestinal disorders) | 44 | 2 | 1
Vomiting (Gastrointestinal disorders) | 93 | 12 | 2
Asthenia (General disorders) | 73 | 12 | 1
Chills (General disorders) | 22 | 3 | 1
Fatigue (General disorders) | 175 | 24 | 0
Oedema peripheral (General disorders) | 48 | 23 | 3
Pyrexia (General disorders) | 29 | 10 | 2
Pneumonia (Infections and infestations) | 11 | 9 | 1
Upper respiratory tract infection (Infections and infestations) | 18 | 11 | 2
Urinary tract infection (Infections and infestations) | 28 | 7 | 4
Overdose (Injury, poisoning and procedural complications) | 39 | 7 | 0
Blood creatinine increased (Investigations) | 22 | 5 | 0
Neutrophil count decreased (Investigations) | 29 | 0 | 0
Platelet count decreased (Investigations) | 26 | 0 | 0
Weight decreased (Investigations) | 42 | 9 | 2
Weight increased (Investigations) | 6 | 8 | 0
Decreased appetite (Metabolism and nutrition disorders) | 101 | 17 | 3
Dehydration (Metabolism and nutrition disorders) | 57 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 23 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 61 | 6 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 58 | 9 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 29 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 12 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 12 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 30 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 10 | 1
Dizziness (Nervous system disorders) | 57 | 12 | 1
Dysgeusia (Nervous system disorders) | 56 | 2 | 0
Headache (Nervous system disorders) | 23 | 4 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 152 | 56 | 6
Anxiety (Psychiatric disorders) | 30 | 4 | 0
Insomnia (Psychiatric disorders) | 53 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 72 | 15 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 76 | 13 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 79 | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 28 | 5 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 | 10 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 105 | 6 | 2
Hypotension (Vascular disorders) | 50 | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (5):
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT02027428/SAP_000.pdf
  • Study Protocol: ABI-007-NSCL-003_protocol_AM1_Redacted 28 October 2014 (2014-10-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02027428/Prot_001.pdf
  • Study Protocol: ABI-007-NSCL-003_protocol_AM2_Redacted.27May2015 (2015-05-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT02027428/Prot_002.pdf
  • Study Protocol: ABI-007-NSCL-003_protocol_AM3_Redacted.13March2017 (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT02027428/Prot_003.pdf
  • Study Protocol: ABI-007-NSCL-003.OriginalProtocolRedacted.27September2013 (2013-09-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT02027428/Prot_004.pdf